CLINICAL TRIAL: NCT05563831
Title: Evaluation Nationale Des Enfants et Adultes Avec Syndromes d'Hypercroissance Dysharmonieuse National Evaluation of Patients With PIK3CA-Related Overgrowth Spectrum (PROS)
Brief Title: National Evaluation of Patients With PIK3CA-Related Overgrowth Spectrum (PROS)
Acronym: COSY
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-09
Record Dates: First submitted 2022-07-28; First posted 2022-10-03 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: PIK3CA-related Overgrowth Spectrum; CLOVES Syndrome; Klippel Trenaunay Syndrome; Megalencephaly; MCAP; Macrodactyly; Vascular Malformations; Lymphatic Malformation; Venous Malformation
Keywords: PIK3CA; Related Overgrowth Syndrome; PIK3CA/AKT/mTOR pathway; clinical diagnosis; Biobank; Patient Stratification
MeSH Terms: conditions — Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi; Klippel-Trenaunay-Weber Syndrome; Megalencephaly; Megalodactyly; Vascular Malformations; Lymphatic Abnormalities; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biopsies and tissues removed during surgical procedures will be stored in the Department of Pathology of Hôpital Necker-Enfants Malades (authorization CODECOH n° DC-2020-3940 de la Plateforme de Resource Biologique de l'Hôpital Necker-Enfants Malades).
  DNA, PBMC and plasma from patients will be stored for further studies. Samples will be stored at the au Centre de Ressources Biologiques de la Structure Fédérative de Recherche Necker (autorisation CODECOH n° DC-2020-3940 du CRB Necker, supervised by Dr. Marie-Alexandra ALYANAKIAN).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: national registry — The investigators will collect demographic, clinical, biological and imaging characteristics of patients with PROS.

SUMMARY:
Overgrowth syndromes are rare genetic disorders defined by tissue hypertrophy that can be either localized or generalized, affecting both latitudinal and longitudinal growth. The genes involved in overgrowth syndromes are not well characterized but mostly concern the PIK3CA/AKT/mTOR pathway, a major actor of cell growth and proliferation. The mutations are not inherited but occurs during embryogenesis leading to somatic mosaicism. Owing to the variability of the clinical presentation, their exact prevalence is yet unknown. In order to answer this question, the investigators team create here the first French national registry on overgrowth syndromes.

DETAILED DESCRIPTION:
Overgrowth syndromes are rare genetic disorders defined by tissue hypertrophy that can be either localized or generalized, affecting both latitudinal and longitudinal growth. The genes involved in overgrowth syndromes are not well characterized but mostly concern the PIK3CA/AKT/mTOR pathway, a major actor of cell growth and proliferation. The mutations are not inherited but occurs during embryogenesis leading to somatic mosaicism. Owing to the variability of the clinical presentation, their exact prevalence is yet unknown. In order to answer this question, the investigators team create here the first French national registry on overgrowth syndromes.

ELIGIBILITY:
Inclusion Criteria:

1. Affiliated to the French healthcare insurance system.
2. Pediatric and adult patients
3. Clinical diagnosis of overgrowth syndrome
4. Written informed consent from adult patients and from both parents of pediatric patients.

Exclusion Criteria:

1. Person subject to a judicial safeguard measure
2. Inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with overgrowth syndrome referred by their doctors or patients who have sent a consultation request to the Reference Center (https://hopital-necker.aphp.fr/contacts-cloves) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of patients with overgrowth syndromes | 5 years
  Clinical and molecular characterization of patients with overgrowth syndromes will be performed.

SECONDARY OUTCOMES:
Prevalence of overgrowth syndromes in France | 5 years
  An estimation of the prevalence of overgrowth syndromes in France will be done
Biobanking of samples derived from patients with overgrowth syndromes | 5 years
  A biobank will be created with biological samples (plasma) collected for research and residual biological samples from patient cares (treatment/diagnosis)
Description of patient cares: mumber of consultations and hospitalizations, number of treatment lines, grouping of patients by type of course (clusters) | 5 years
  An analysis of care trajectories will be performed. These data will be collected from health insurance databases for patients with overgrowth syndromes.
Economic evaluation of cares for patients with overgrowth syndromes: cost of care, per period and cumulative. | 5 years
  SDNS data will be used to estimate care costs per year for patients with overgrowth syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Canaud, MD,PHD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Translational medicine and Targeted therapies unit, Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canaud G, Hammill AM, Adams D, Vikkula M, Keppler-Noreuil KM. A review of mechanisms of disease across PIK3CA-related disorders with vascular manifestations. Orphanet J Rare Dis. 2021 Jul 8;16(1):306. doi: 10.1186/s13023-021-01929-8. PMID 34238334
- [Background] Morin G, Canaud G. Treatment strategies for mosaic overgrowth syndromes of the PI3K-AKT-mTOR pathway. Br Med Bull. 2021 Dec 16;140(1):36-49. doi: 10.1093/bmb/ldab023. PMID 34530449
- [Background] Delestre F, Venot Q, Bayard C, Fraissenon A, Ladraa S, Hoguin C, Chapelle C, Yamaguchi J, Cassaca R, Zerbib L, Magassa S, Morin G, Asnafi V, Villarese P, Kaltenbach S, Fraitag S, Duong JP, Broissand C, Boccara O, Soupre V, Bonnotte B, Chopinet C, Mirault T, Legendre C, Guibaud L, Canaud G. Alpelisib administration reduced lymphatic malformations in a mouse model and in patients. Sci Transl Med. 2021 Oct 6;13(614):eabg0809. doi: 10.1126/scitranslmed.abg0809. Epub 2021 Oct 6. PMID 34613809
- [Background] Morin G, Degrugillier-Chopinet C, Vincent M, Fraissenon A, Aubert H, Chapelle C, Hoguin C, Dubos F, Catteau B, Petit F, Mezel A, Domanski O, Herbreteau G, Alesandrini M, Boddaert N, Boutry N, Broissand C, Han TK, Branle F, Sarnacki S, Blanc T, Guibaud L, Canaud G. Treatment of two infants with PIK3CA-related overgrowth spectrum by alpelisib. J Exp Med. 2022 Mar 7;219(3):e20212148. doi: 10.1084/jem.20212148. Epub 2022 Jan 26. PMID 35080595
- [Result] Venot Q, Blanc T, Rabia SH, Berteloot L, Ladraa S, Duong JP, Blanc E, Johnson SC, Hoguin C, Boccara O, Sarnacki S, Boddaert N, Pannier S, Martinez F, Magassa S, Yamaguchi J, Knebelmann B, Merville P, Grenier N, Joly D, Cormier-Daire V, Michot C, Bole-Feysot C, Picard A, Soupre V, Lyonnet S, Sadoine J, Slimani L, Chaussain C, Laroche-Raynaud C, Guibaud L, Broissand C, Amiel J, Legendre C, Terzi F, Canaud G. Targeted therapy in patients with PIK3CA-related overgrowth syndrome. Nature. 2018 Jun;558(7711):540-546. doi: 10.1038/s41586-018-0217-9. Epub 2018 Jun 13. PMID 29899452
- [Result] Manning BD, Toker A. AKT/PKB Signaling: Navigating the Network. Cell. 2017 Apr 20;169(3):381-405. doi: 10.1016/j.cell.2017.04.001. PMID 28431241